CLINICAL TRIAL: NCT01645995
Title: The Impact of Reformulated Product Consumption on Energy and Nutrient Intake, Body Composition, Vascular Function and Plasma Lipid and Glucose Concentrations
Brief Title: The Impact of Reformulated Foods on Cardiovascular Risk Factors
Acronym: REFORM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Responsible Party: Principal Investigator, Julie Lovegrove, Professor of Metabolic Nutrition, University of Reading
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 12/03
Record Dates: First submitted 2012-07-18; First posted 2012-07-20 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Type 2 Diabetes Mellitus; Cardiovascular Disease; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Reformulated products (Experimental): Subjects were asked to supplement their habitual diet with reformulated sugar-reduced products for 8 weeks. Subjects were provided with reformulated beverages, sauces, condiments and snacks. They were asked to consume a minimum of 1 drink + 1 food portion intervention supplement daily, in exchange for habitually eaten equivalent foods.
  Interventions: Dietary Supplement: Reformulated products
- Conventional products (Experimental): Subjects were asked to supplement their habitual diet with conventional sugar products for 8 weeks. Subjects were provided with conventional beverages, sauces, condiments and snacks. They were asked to consume a minimum of 1 drink + 1 food portion intervention supplement daily, in exchange for habitually eaten equivalent foods.
  Interventions: Dietary Supplement: Conventional products

INTERVENTIONS:
Dietary Supplement: Reformulated products — Subjects were asked to supplement their habitual diet with reformulated sugar-reduced products for 8 weeks. Subjects were provided with reformulated beverages, sauces, condiments and snacks. They were asked to consume a minimum of 1 drink + 1 food portion intervention supplement daily, in exchange for habitually eaten equivalent foods.
  Other Names: REF
  Arms: Reformulated products
Dietary Supplement: Conventional products — Subjects were asked to supplement their habitual diet with conventional sugar products for 8 weeks. Subjects were provided with conventional beverages, sauces, condiments and snacks. They were asked to consume a minimum of 1 drink + 1 food portion intervention supplement daily, in exchange for habitually eaten equivalent foods.
  Other Names: CON
  Arms: Conventional products

SUMMARY:
Specific policies on obesity reduction often include a recommendation to reduce sugar consumption as a means of lowering overall caloric intake. Reformulating processed foods (e.g. sugary products) is considered one of the key options for improving population diet. The implications of regular consumption of reformulated products are not fully understood. Previous studies have demonstrated that dietary compensation is common, although the extent is not fully elucidated. In addition to the perceived impact of sugar consumption on weight control, high sugar intake, specifically sucrose and fructose, has been implicated in the increase of plasma lipids and markers of insulin resistance. However to date no randomised controlled study has investigated whether the consumption of reformulated low sugar products as components of a habitual diet have a significant impact on plasma lipid, insulin or glucose concentrations within a free-living, non-diseased population. It is hypothesised that exchange of reformulated, low sugar food products for habitually consumed foods will result in dietary compensation and minimal weight change compared with unmodified products and will have little impact on plasma glucose, insulin and lipid levels.

ELIGIBILITY:
Inclusion Criteria:

* Age: 20 - 49 years
* BMI 18.5 - 30 kg/m2
* Plasma glucose <7 mmol/l (Not diagnosed with diabetes)
* Plasma cholesterol <7 mmol/l
* Plasma TAG <2.3 mmol/l
* Normal liver and kidney function
* Haemoglobin (>110 g/l women; 140g/dl men)

Exclusion Criteria:

* Having suffered a myocardial infarction/stroke in the past 12 months
* diabetic (diagnosed or fasting glucose > 7 mmol/l)
* Smoking
* On drug treatment for hyperlipidaemia, hypertension, inflammation or hypercoagulation
* Suffering from renal or bowel disease or have a history of choleostatic liver or pancreatitis
* Excessive alcohol consumption
* History of alcohol abuse
* Following a reducing diet or vegan diet
* Taking any fish oil, fatty acid or vitamin and mineral supplements
* Participating in intensive aerobic activity for > 20 minutes 3 times per week
* Food allergies
* Anti-inflammatory usage

Ages: 20 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2012-03; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Changes in body weight and body composition | 20 weeks. Baseline and week 8 assessments for two dietary intervention arms

SECONDARY OUTCOMES:
Changes in energy and nutrient intake | 20 weeks. Run-in period and week 7 assessments for two dietary intervention arms
Changes in appetite and mood ratings | 20 weeks. Run-in period and week 7 assessments for two dietary intervention arms
  Subjective sensations of appetite and mood by visual analogue scale
Changes in physical activity levels | 20 weeks. Run-in period and week 7 assessments for two dietary intervention arms
  Measured by accelerometry
Changes in fasting plasma lipid, insulin and glucose concentrations | 20 weeks. Baseline and week 8 assessments for two dietary intervention arms
Changes in vascular stiffness by pulse wave analysis (PWA) and digital volume pulse (DVP) | 20 weeks. Baseline and week 8 assessments for two dietary intervention arms
Changes in cardiovascular risk factors (blood pressure, inflammatory markers) | 20 weeks. Baseline and week 8 assessments for two dietary intervention arms

CONTACTS AND LOCATIONS:
Overall Officials: Prof Julie A Lovegrove, BSc, PhD, RNutr, Principal Investigator — University of Reading
Locations (1):
- Department of Food and Nutritional Sciences, University of Reading, Reading, Berks, United Kingdom

REFERENCES:
- [Result] Reid M, Hammersley R, Duffy M. Effects of sucrose drinks on macronutrient intake, body weight, and mood state in overweight women over 4 weeks. Appetite. 2010 Aug;55(1):130-6. doi: 10.1016/j.appet.2010.05.001. Epub 2010 May 12. PMID 20470840
- [Result] Reid M, Hammersley R, Hill AJ, Skidmore P. Long-term dietary compensation for added sugar: effects of supplementary sucrose drinks over a 4-week period. Br J Nutr. 2007 Jan;97(1):193-203. doi: 10.1017/S0007114507252705. PMID 17217576